CLINICAL TRIAL: NCT03920384
Title: Improving Psychological Therapy for Psychosis: A Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203489
Record Dates: First submitted 2019-02-26; First posted 2019-04-18 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-04

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Randomised case series
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental therapy arm (Experimental): 16 (minimum 4, maximum 20) sessions of therapy for psychosis including new therapeutic ingredients
  Interventions: Behavioral: Experimental intervention arm
- Standard Psychological Therapy for Psychosis (Active Comparator): 16 (minimum 4 maximum 20) sessions of standard psychological therapy for psychosis.
  Interventions: Behavioral: Active control arm

INTERVENTIONS:
Behavioral: Experimental intervention arm — Psychological therapy for psychosis with new therapy components
  Arms: Experimental therapy arm
Behavioral: Active control arm — Standard psychological therapy for psychosis without new therapy components
  Arms: Standard Psychological Therapy for Psychosis

SUMMARY:
Standard psychological therapy for psychosis (Cognitive Behavioural Therapy) is made up of different 'ingredients', also called treatment components. In therapy, different treatment components can be included or excluded depending on the needs of the individual. In this study, the investigators want to find out if standard psychological therapy for psychosis can be improved by including new treatment components. Therefore, participants in this study will be offered psychological therapy for psychosis with new treatment components included or standard psychological therapy for psychosis without new treatment components included. Which of these two options participants are offered will be decided by chance, and during the study neither the study participants nor the researcher will know which of these two variations of psychological therapy are given. Researchers call this a randomized double-blind study. The investigators are aiming to use the results from this study to guide the improvement of psychological therapies for psychosis.

DETAILED DESCRIPTION:
Individuals with psychosis often experience delusions, hallucinations and disorganised thinking. Clinicians call these 'positive symptoms' as they are seen as an addition to regular functioning. Psychosis can also lead to loss of some functions such as lower motivation and decreased interest in activities; these are called 'negative symptoms'. Even though most people receive medication for psychosis, psychological therapies such as Cognitive Behavioural Therapy for psychosis (CBTp) are also important in terms of managing symptoms and increasing well-being. Standard CBTp is made up of different treatment components and in therapy, different treatment components can be included or excluded depending on the needs of the individual. In this study the investigators are looking to identify treatment components that are beneficial to CBTp. In particular, the aim is to test whether adding some newly developed treatment components to CBTp can lead to additional benefits to patients, in terms of reducing unhelpful thinking styles. This will be done through a double-blind randomized case-series design, where participants will either receive standard CBTp or standard CBTp with added treatment components.

Four weeks before the intervention starts, throughout therapy, as well as four weeks after therapy, participants will complete weekly questionnaires to assess symptoms and thinking patterns. This will allow the researcher to measure weekly changes before, during and after the therapy. Additional questionnaires and interviews as well as computer tasks will also be completed before the therapy starts (baseline), mid-therapy and post-therapy to gain more insight into changes in mood, quality of life, thinking patterns and symptoms. In addition, to study the long-term effect of the intervention, participants will be asked to complete a follow-up assessment session 12 weeks after the therapy is completed. Participants and clinicians will also be given the opportunity to give feedback on their experience of having received/delivered the therapy. This will be done through an interview with the researcher, and will give us further insight into how future therapies for psychosis might be improved, both from a clinician and patient perspective.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 16 or over
* Are competent and willing to provide written, informed consent
* Are experiencing delusions (A score of ≥3 on PANSS item P1, P5 or P6)

Exclusion Criteria:

* Significant developmental disability
* Currently receiving or have received CBTp in the last 6 months
* Significant difficulty with the English language

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Session by session change in positive symptoms as measured by the The Psychotic Symptom Rating Scales (PSYRATS, Haddock et al.,1999). | Administered weekly 4 weeks prior to therapy start, weekly after each therapy session (maximum 20 sessions) and weekly for 4 weeks after therapy intervention has been completed as well as 12 weeks follow-up after intervention completion.
  The PSYRATS is a widely used measure including 17 items assessing different dimensions of delusions and auditory hallucinations that include distress, loudness, conviction, frequency, disruption to life and preoccupation. Each dimension is rated on a 0-4 point scale, with scores on the auditory hallucination subscale (11 items) ranging from 0-44 and scores on the delusion subscale (6 items) ranging from 0-24. Higher scores indicate greater symptom severity.
Session by session change in cognitive biases measured by Davos Assessment of Cognitive Biases Scales (DACOBS: van der Gaag et al., 2013). | Assessed weekly for 4 weeks prior to therapy start, weekly after each therapy session (maximum 20 sessions) and weekly for 4 weeks after therapy intervention has been completed.
  This scale consists of 42 statements relating to seven (six-item) subscales; 1) Jumping to conclusions bias 2) Belief inflexibility bias 3) Attention to threat bias 4) External attribution bias 5) Social cognition problems 6) Subjective cognitive problems and 7) Safety behaviours. Respondents score each statement using a 7-point rating scale, ranging from 'totally disagree' (1) to 'totally agree' (7). For the session-by session data, the subscales Jumping to conclusions, Belief Inflexibility Bias and External Attribution bias subscales will be administered. Each cognitive bias subscale obtains a score from 7-42, with a higher score indicating higher propensity towards a cognitive bias.

SECONDARY OUTCOMES:
Jumping to conclusions task (Garety et al., 1991; Moritz et al., 2010). | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  A computerised task where participants are presented with two lakes of coloured fish in opposing ratios (e.g. Lake A 80% red 20% green, Lake B 80% green 20% red). The participant is told that the fisherman will fish from one of these lakes only (but which lake is unknown). After each "catch" the participant is asked to make 2 judgements: 1) probability that the fish is caught from lake A or B and 2) Whether they are ready to make a decision on what lake the fish is caught from. This task measures participants tendency to jump to conclusions.
Bias Against Disconfirmatory Evidence (BADE) task (Woodward et al., 2006) | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  A computerised version of the BADE task will be employed. In this task, participants will be presented a series of with delusion-neutral scenarios. For each scenario they will be asked to rate the plausibility of 4 interpretations each scenario will have a one "true" interpretation two "lure" interpretation and one "absurd" interpretation. After making their ratings, participants will be presented with additional scenario descriptions, which will provide further information, and participants will be allowed to adjust their ratings if necessary
Positive and Negative Syndrome Scale (PANSS; Kay et al., 1987) | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  PANSS is a structured clinical interview that estimates symptom severity for people with schizophrenia and psychosis. The scale consists of 30 items measuring positive (P1-P7), negative (N1-N7) and general (G1-G16) symptom severity. Each of the items is scored on a 1-7 point scale ranging from absent (1) to extreme (7). Total scores range from 30-210, with higher scores indicating greater symptom severity.
Internalized Stigma of Mental Illness Scale (ISMI; Ritsher et al., 2003) | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  This is a 29-item questionnaire that assesses subjective levels of self-stigma. Participants are asked to rate the extent to which they agree with a set of statements on a 1-4 point scale scale ranging from strongly disagree (1) to strongly agree (4). Items add up to 5 subscales, including: alienation, stereotype endorsement, discrimination experience, social withdrawal and stigma resistance. Scores for subscales and total scores are calculated by adding the item scores and dividing by total number of answered items, with higher scores indicating higher internalized stigma.
Calgary Depression Scale for Schizophrenia (CDSS; Addington et al., 1990). | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  Measures depressive symptoms in schizophrenia. The scale consists of a structured interview with nine questions, and are scored on a 0-3 scale ranging from absent (0) to severe (3). Total score range 0-27 with higher scores indicating higher severity of depressive symptoms.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-18; Ritsner et al., 2005). | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  An 18-item self-administered questionnaire designed to assess quality of life in patients with psychotic and mood disorders. It is a self-administered scale where participants are asked to rate questions on a 1-5 scale, ranging from "not at all or never" (1) to "Frequently or all of the time" (5). Total scores range from 18-90 and a higher score indicates higher a quality of life.
The Global Assessment of Functioning (GAF; American Psychological Association, APA, 1987) | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  The GAF scale is a rating scale for assessing a person's psychological, social and occupational functioning. The scale total ranges from 1-100, where a lower score indicates a more severe illness in terms of symptoms and social functioning.
The Reflective Function Questionnaire (RFQ short version: Fonagy & Ghinai (unpublished manuscript) | Administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  8-item scale to assess mentalising capacity in adults. Total scores range from 8-42. The RFQ-8 contains median scored items where scores in the middle ("partly agree" or "partly disagree") get high scores, while responses in the extreme ends of the scale reflect poor mentalising capacity.
Change in cognitive biases measured by Davos Assessment of Cognitive Biases Scales (DACOBS: van der Gaag et al., 2013). | Full scale administered at 6 study assessment points: Pre-baseline (4 weeks prior to therapy start), Baseline (pre-therapy start), Post therapy session 8, Post-Therapy completion (maximun 20 sessions), as well as weeks 4 and 12 post therapy completion.
  This scale consists of 42 statements relating to seven (six-item) subscales; 1) Jumping to conclusions bias 2) Belief Inflexibility bias 3) Attention to threat bias 4) External attribution bias 5) Social cognition problems 6) Subjective cognitive problems and 7) Safety behaviours. Respondents score each statement using a 7- point rating scale, ranging from 'totally disagree' (1) to 'totally agree' (7). Each cognitive bias subscale obtains a score from 7-42, with a higher score indicating higher propensity towards a cognitive bias.

OTHER OUTCOMES:
Qualitative questions post-intervention | Interview will be done after participants have completed the therapy intervention (an average of 6 months after study commencement). Trial therapists will be interviewed once their study interventions are completed with trial participants.
  A semi-structured interview will be conducted with both clinicians and participants after the intervention. This interview will centre around the themes of subjective experiences of the therapy, subjective experiences of change, mechanisms of change and useful versus less useful aspects of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Eliasson, Principal Investigator — University of Edinburgh
Locations (1):
- Lothian NHS Board, Edinburgh, Scotland, United Kingdom